CLINICAL TRIAL: NCT01643356
Title: Interventions to Reduce Excess Weight Gain in Pregnancy in Overweight and Obese Mothers
Brief Title: Interventions to Reduce Excess Weight Gain in Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Responsible Party: Principal Investigator, Susan Roberts, Director, Energy Metabolism Laboratory, Tufts University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 10203 Tufts
Record Dates: First submitted 2012-07-16; First posted 2012-07-18 (Estimated); Last update posted 2016-05-10 (Estimated); Status verified 2016-05

CONDITIONS: Overweight and Obesity; Pregnancy
Keywords: weight; pregnancy; behavioral intervention; obesity
MeSH Terms: conditions — Overweight; Obesity; Body Weight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Fiber Cereal (Active Comparator): Women assigned to this arm will receive the group based behavioral intervention plus the recommendation to consume provided high fiber cereal to manage hunger.
  Interventions: Behavioral: Intervention to reduce excess weight gain during pregnancy
- Control Group (No Intervention): Women assigned to this arm of the study will receive routine clinical care and no additional interventions.
- Resistant Starch (Active Comparator): Women assigned to this arm will receive the group based behavioral intervention plus the recommendation to consume provided resistant starch to control hunger
  Interventions: Behavioral: Intervention to reduce excess weight gain during pregnancy

INTERVENTIONS:
Behavioral: Intervention to reduce excess weight gain during pregnancy — Intervention includes meetings with a nutrition counselor and/or psychologist where individualized eating plans will be developed and reviewed, and regular group meetings during which information about healthy eating for weight management will be discussed.
  Arms: Fiber Cereal; Resistant Starch

SUMMARY:
The study will use a comprehensive behavioral intervention adapted for pregnant women to change dietary intake, eating behavior and physical activity. The central hypothesis of this study is that the intervention will reduce excess gestational weight gain and achieve clinical and metabolic benefits in obese and overweight pregnant women and their infants over the first year of life.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-45 years
* In first trimester of pregnancy
* Must be willing to not join any other weight control program while in the study
* BMI of 25-40 kg/m2
* Willingness and ability to attend support group meetings either in person or via web
* Must be able to read, speak, and understand English

Exclusion Criteria:

* Carrying multiple fetuses
* Gestational diabetes mellitus at study entry
* Type 2 diabetes mellitus or blood glucose >125 mg/dl at screening
* Self reported current substance abuse
* Current smoking
* Alchol consumption of more than 1 drink per day
* Preexisting medical conditions (includes bariatric surgery) or use of medications that would impact study involvement or outcomes testing
* Eating disorder in the past 2 years
* Depression or diagnosis of bipolar disorder
* Concurrent participation in any other research study that would impact participation in this investigation

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2012-07; Primary Completion 2014-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Maternal and Infant Body Weight Change | From first trimester through 1 year post-partum
  * Maternal non-fasting weight measured at all prenatal clinic and study visits.
  * Infant weight measured at birth and all pediatric clinic visits through 1 year.

SECONDARY OUTCOMES:
Infant Outcomes | From birth through first year
  * Body composition (i.e. length, head circumference, skinfold thickness, waist circumference) changes through the first year.
  * Characteristics at birth including Apgar score, gestational age.
  * Dietary intake and food preferences at 1 year.
Maternal and Perinatal Outcomes | First trimester through 1 year post-partum
  * Rates of cesarean delivery, gestational hypertension/preeclampsia, preterm birth, birth complications.
  * Fasting blood glucose and insulin concentrations throughout pregnancy.
  * Body composition and energy requirements at baseline and 24-28 weeks of pregnancy.
  * Total energy expenditure at 24-28 weeks of pregnancy.
  * Rate of breastfeeding and breastfeeding practices at 1, 3, 6, and 12 months post-partum.

CONTACTS AND LOCATIONS:
Overall Officials: Susan B Roberts, Ph.D., Principal Investigator — Tufts University
Locations (2):
- United States (2):
  - Tufts Medical Center, Boston, Massachusetts
  - Tufts University Human Nutrition Research Center on Aging, Boston, Massachusetts